CLINICAL TRIAL: NCT06084845
Title: Phase II Trial of Xevinapant and Chemoradiotherapy in Adjuvant Treatment for Patients With Head and Neck Squamous Cell Carcinoma With High Risk Pathologic Features
Brief Title: Testing the Addition of an Investigational Drug, Xevinapant, to Usual Radiation Therapy Plus Cisplatin/Carboplatin for Patients With Head and Neck Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A phase III trial of the investigational agent failed to pass futility boundaries at interim analysis
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA3222; NCI-2023-06677 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA3222 (Other: ECOG-ACRIN Cancer Research Group); EA3222 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Specimen Handling; Carboplatin; X-Rays; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (chemoradiation) (Active Comparator): Patients receive cisplatin or carboplatin IV over 30-60 minutes QW for 6 doses with concurrent IMRT and IGRT five days a week for 30-33 fractions in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, PET-CT, and/or chest x-ray during screening and follow-up. Patients may also undergo blood sample collection during follow-up.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Chest Radiography; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Arm B (chemoradiation, xevinapant) (Experimental): Patients receive cisplatin or carboplatin IV over 30-60 minutes QW for 6 doses with concurrent IMRT and IGRT five days a week for 30-33 fractions in the absence of disease progression or unacceptable toxicity. Patients also receive xevinapant PO on days 1-14 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, PET-CT, and/or chest x-ray during screening and follow-up. Patients may also undergo blood sample collection during follow-up.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Chest Radiography; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Xevinapant

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT and/or PET-CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Radiation: Image Guided Radiation Therapy — Undergo IGRT
  Other Names: IGRT; image-guided radiation therapy; Image-Guided Radiotherapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET-CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Xevinapant — Given PO
  Other Names: AT-406; D1143; Debio 1143; Debio-1143; Debio1143; IAPs Antagonist Debio 1143; IAPs Inhibitor Debio 1143; Pyrrolo(1,2-a)(1,5)diazocine-8-carboxamide, n-((1,1'-biphenyl)-2-ylmethyl)decahydro-5-(((2s)-2-(methylamino)-1-oxopropyl)amino)-3-(3-methyl-1-oxobutyl)-6-oxo-, (5s,8s,10ar); Second Mitochondrial-derived Activator of Caspases Mimetic Debio 1143; SM-406; SMAC Mimetic Debio 1143
  Arms: Arm B (chemoradiation, xevinapant)

SUMMARY:
This phase II trial compares the effect of usual radiation therapy with cisplatin/carboplatin (chemoradiation) to the addition of xevinapant with chemoradiation in patients with head and neck cancer. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of cancer cells. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of cancer cells. Xevinapant is a first-in-class antagonist of inhibitor of apoptosis (programmed cell death) proteins (IAPs), which leads to tumor cell death and enhances tumor cell sensitivity to chemotherapy and radiotherapy. Giving xevinapant with chemoradiation may be more effective in preventing head and neck cancer from growing or spreading than chemoradiation alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether adding xevinapant to post-operative adjuvant treatment with cisplatin + radiation followed by xevinapant monotherapy in patients with surgically resected head and neck squamous cell carcinoma (HNSCC) who have extra-nodal extension (ENE) and/or positive margins will improve the disease-free survival (DFS).

SECONDARY OBJECTIVES:

I. To evaluate the following endpoints: Overall Survival (OS), rates of distant metastasis (DM), local regional control (LRR).

II. To assess safety and tolerability of treatment intensification.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive cisplatin or carboplatin intravenously (IV) over 30-60 minutes once a week (QW) for 6 doses with concurrent intensity-modulated radiation therapy (IMRT) and image guided radiation therapy (IGRT) five days a week for 30-33 fractions in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET)-CT, and/or chest x-ray during screening and follow-up. Patients may also undergo blood sample collection during follow-up.

ARM B: Patients receive cisplatin or carboplatin IV over 30-60 minutes QW for 6 doses with concurrent IMRT and IGRT five days a week for 30-33 fractions in the absence of disease progression or unacceptable toxicity. Patients also receive xevinapant orally (PO) on days 1-14 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, PET-CT, and/or chest x-ray during screening and follow-up. Patients may also undergo blood sample collection during follow-up.

Upon completion of study treatment, patients are followed up at 30 days and every 6 months if patient is < 3 years from randomization and every 12 months if patient is 3-5 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age
* Patient must have stage III or IVA or IVB HPV-negative squamous cell carcinoma of the head and neck (HNSCC) by American Joint Committee on Cancer (AJCC) Cancer Staging Manual, 8th edition criteria
* Patient must have undergone gross total surgical resection of high-risk oral cavity, oropharynx (p16 negative), larynx, or hypopharynx within 63 days prior to randomization
* Patient must have evidence of high-risk features on final postoperative pathology including positive margins (R1) and/or extranodal extension. Patients with gross residual disease are not eligible
* Patient must have tumor origin site in the oral cavity, oropharynx, larynx, or hypopharynx
* Patient must have received no prior treatment for HNSCC with the exception of curative intent surgical resection
* Patient must have imaging consisting of CT of the head, neck and chest within 10 weeks prior to randomization to confirm there is no evidence of disease
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and continue contraception measures for 6 months after the last dose of cisplatin or carboplatin and for 3 months after the last dose of xevinapant. Patient must not breast-feed while on protocol treatment and for one month after the last dose of any protocol treatment. Patient must not donate sperm while on protocol treatment
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* White blood cell (WBC) ≥ 3,000/mcL (obtained ≤ 14 days prior to protocol randomization)
* Absolute neutrophil count (ANC) ≥ 1,500/mcL (obtained ≤ 14 days prior to protocol randomization)
* Platelets ≥ 100,000/mcL (obtained ≤ 14 days prior to protocol randomization)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (obtained ≤ 14 days prior to protocol randomization)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) ≤ 3.0 × institutional ULN (obtained ≤ 14 days prior to protocol randomization)
* Creatinine clearance ≥ 60 mL/min (estimated using Cockcroft-Gault method or measured) (obtained ≤ 14 days prior to protocol randomization)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial. Patients with HIV must have viral load monitored as clinically indicated
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with non-compensated or symptomatic liver cirrhosis (Child-Pugh score: B or C) are not eligible
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. Patients with non-compensated or symptomatic liver cirrhosis (Child-Pugh score: B or C) are not eligible
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patient must not have had a live-attenuated vaccine within 30 days prior to randomization
* Patient must not have a known gastrointestinal disorder with clinically established malabsorption syndrome and major gastrointestinal surgery that may limit oral absorption
* Patient must not have taken any agents on the prohibited medication list within 14 days prior to randomization or require any of these agents for ongoing treatment while on protocol treatment
* Patient must not have active, uncontrolled inflammatory disease (including rheumatoid arthritis, systemic lupus erythematosus, Sjögren syndrome, severe extensive psoriasis, and other autoimmune diseases) requiring ongoing treatment with anti-tumor necrosis factor (TNF) medication
* Patient must have had a pre-surgical or other baseline electrocardiogram (EKG) report within 6 months prior to randomization indicating a corrected QT (QTc) using Fridericia's formula (QTcF) interval < 450 ms for males and < 470 ms for females
* Patient must not be on any concomitant medication known to prolong the QTcF interval that cannot be discontinued or replaced by safe alternative medication within 7 days prior to randomization
* Patient must not have a known allergy to xevinapant, cisplatin, carboplatin, other platinum-based agent or any excipient known to be present in any of these products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-12 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | From the date of randomization to the date of recurrence, second primary tumor from the head and neck region, or death, assessed at 2 years
  Assuming an exponential distribution for DFS, this hypothesis corresponds to an increase in the 2-year DFS rate from 55% (assumed rate in the control arm) to 70%. Full information required will be a total of 100 DFS events. An intention to treat analysis including all randomized patients will be used. Kaplan-Meier estimates will be used to estimate the DFS distributions. A log-rank test with a one-sided 10% type I error will be used for the comparison between the arms.

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death from any cause, assessed at 2 years
  Assuming a 2-year OS rate of 69% in the control arm, maintaining a one-sided significance level of 10%, there is 80% power to detect a hazard ratio of 1.66, for the comparison of control arm versus experimental arm. Assuming an exponential distribution for OS, this hypothesis corresponds to an increase in the 2-year OS rate from 69% to 80%. Full information will be a total of 72 OS events.
Incidence of adverse events | Up to 30 days post completion of treatment
  All treated patients will be evaluated for toxicity (using the Common Terminology Criteria for Adverse Events) regardless of eligibility. Toxicity will be examined by arm and compared using the Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Heath D Skinner, Principal Investigator — ECOG-ACRIN Cancer Research Group